CLINICAL TRIAL: NCT03903471
Title: Comparion of 22G-ProCore and 22G-Standard Needle in Diagnosis of Lymphadenopathy Via EBUS-TBNA: A Prospective, Single-center, Randomized Controlled Clinical Trial
Brief Title: 22G-ProCore vs 22G-Standard Needle in Diagnosis of Lymphadenopathy by EBUS-TBNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiayuan Sun (Other)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy and Interventional Pulmonology, Shanghai Chest Hospital, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHCHE201901
Record Dates: First submitted 2019-03-31; First posted 2019-04-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Lymph Node Disease
Keywords: ProCore; Mediastinal and Hilar Lymphadenopathy; EBUS-TBNA; Diagnostic Yield; Quality of Specimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 22G-ProCore Group (Experimental): The experimental group with 22G-ProCore needle is expected to enroll 300 patients. The 22G-ProCore needle has a 1.5mm long groove 2.5mm above the needle tip, which is expected to have the advantage of taking more biopsy tissues than the 22G-Standard needle.
  Interventions: Device: 22G-ProCore Endobronchial Ultrasound Needle
- 22G-Standard Group (Active Comparator): The control group of 22G-Standard needle is expected to include 300 patients, and there is no groove above the needle tip compared with 22G-ProCore needle.
  Interventions: Device: 22G-Standard Endobronchial Ultrasound Needle

INTERVENTIONS:
Device: 22G-ProCore Endobronchial Ultrasound Needle — EchoTip Procore® Endobronchial HD Ultrasound Biopsy Needle, COOK
  Arms: 22G-ProCore Group
Device: 22G-Standard Endobronchial Ultrasound Needle — EchoTip® Ultra Endobronchial High Definition Ultrasound Needle, COOK
  Arms: 22G-Standard Group

SUMMARY:
The aim of this study is to compare the performance of 22G-ProCore and 22G-Standard needle in diagnosis of mediastinal and hilar lymphadenopathy via EBUS-TBNA with the purpose to explore the optimal technique for obtaining diagnostic material.

DETAILED DESCRIPTION:
EBUS-TBNA is an important minimally invasive tool for the diagnosis of mediastinal and hilar lymphadenopathy. The investigators will explore the performance of two kinds of needles and different methods to obtain tissues via EBUS-TBNA in the study. The study is designed as a prospective, single-center, randomized controlled trial, 600 patients will be expected to enroll in the study and randomly assigned to two groups, the 22G-ProCore group and the 22G-Standard group. The primary aim is to compare the diagnostic yields of the two types of needles. The secondary endpoint is to assess the quality of histologic specimen. Meanwhile, stylet slow-pull or negative suction techniques and different agitations (10, 20, 30 times) that each pass includes will be evaluated in the study as well.

ELIGIBILITY:
Inclusion Criteria:

1. Imaging examination indicates enlarged intrathoracic lymph nodes need pathological diagnosis (any lymph node has a short diameter > 1 cm in CT or PET-CT SUV value > 2.5).
2. Accessible mediastinal and hilar lymphadenopathy to EBUS-TBNA.
3. Inform consent signed.

Exclusion Criteria:

1. Contraindications of EBUS-TBNA. Such as use of anticoagulant therapy or presence of a coagulopathy (platelet count < 50000 or INR > 1.5).
2. Severe cardiopulmonary dysfunction and other indications that can't tolerate bronchoscopy.
3. Life expectancy less than 6 months.
4. Uncooperative patients.
5. Patients representing vulnerable populations (prisoners, pregnant women, etc).
6. Researchers consider it inappropriate to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-08 (Estimated); Primary Completion 2023-10-08 (Estimated); Study Completion 2023-10-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of 22G-ProCore needle | up to 6 months
  Diagnostic yield is defined as percentage of specimens in which diagnostic material is obtained.
Diagnostic yield of 22G-Standard needle | up to 6 months
  Diagnostic yield is defined as percentage of specimens in which diagnostic material is obtained.

SECONDARY OUTCOMES:
The quality of histologic specimen used by 22G-ProCore needle | up to 6 months
  The number and ratio of cellularity, blood contamination, and core-tissue acquisition.
The quality of histologic specimen used by 22G-Standard needle | up to 6 months
  The number and ratio of cellularity, blood contamination, and core-tissue acquisition.

OTHER OUTCOMES:
Diagnostic yield of aspiration techniques | up to 6 months
  Conventional EBUS-TBNA procedures involve use of 10mL negative suction aspiration techniques. A new aspiration method, the stylet slow-pull technique, involves slow withdrawal of the needle stylet to create minimum negative pressure.
Diagnostic yield of different agitations | up to 6 months
  Agitation means needle moving 10 or 20 or 30 times back and forth in lymph nodes per pass.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stamatis G. Staging of lung cancer: the role of noninvasive, minimally invasive and invasive techniques. Eur Respir J. 2015 Aug;46(2):521-31. doi: 10.1183/09031936.00126714. Epub 2015 May 14. PMID 25976686
- [Background] Sun J, Zhang J, Zhao H, Shen J, Gu A, Han B. Role of endobronchial ultrasound-guided transbronchial needle aspiration in the diagnosis of bronchogenic carcinoma: Experience of a single institution in China. Thorac Cancer. 2010 May;1(1):28-34. doi: 10.1111/j.1759-7714.2010.00010.x. PMID 27755785
- [Background] Sun J, Teng J, Yang H, Li Z, Zhang J, Zhao H, Garfield DH, Han B. Endobronchial ultrasound-guided transbronchial needle aspiration in diagnosing intrathoracic tuberculosis. Ann Thorac Surg. 2013 Dec;96(6):2021-7. doi: 10.1016/j.athoracsur.2013.07.005. Epub 2013 Sep 12. PMID 24035300
- [Background] Sun J, Yang H, Teng J, Zhang J, Zhao H, Garfield DH, Han B. Determining factors in diagnosing pulmonary sarcoidosis by endobronchial ultrasound-guided transbronchial needle aspiration. Ann Thorac Surg. 2015 Feb;99(2):441-5. doi: 10.1016/j.athoracsur.2014.09.029. Epub 2014 Dec 12. PMID 25497069
- [Background] Yang H, Wang S, Teng J, Han B, Sun J. Utility of endobronchial ultrasound-guided transbronchial needle aspiration in diagnosing non-specific inflammatory intrathorcacic lymphadenitis. Clin Respir J. 2018 Feb;12(2):691-698. doi: 10.1111/crj.12580. Epub 2016 Nov 23. PMID 27882677